CLINICAL TRIAL: NCT07171671
Title: The Effectiveness of Manual Therapy Applications in Individuals With Rheumatoid Arthritis Who Have Temporomandibular Joint Dysfunction
Brief Title: Treatment in Individuals With Rheumatoid Arthritis Who Have Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, director, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hakanpolat4
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Rheumatic Diseases; Temporomandibular Joint Dysfunction; Manuel Therapy
Keywords: Rheumatoid arthritis; Temporomandibular joint dysfunction; Manual therapy; Pain
MeSH Terms: conditions — Rheumatic Diseases; Temporomandibular Joint Disorders; Arthritis, Rheumatoid; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial Mobilisation (Experimental): Myofascial mobilisation treatment was carried out in three stages. In these stages, trigger point therapy was first applied, followed by myofascial release and finally the muscle energy technique for the masticatory muscles. The procedures were performed twice a week for six weeks. The sessions lasted an average of 30 minutes.
  Interventions: Other: exercises
- Joint mobilisation group (Experimental): Joint mobilisation treatment was carried out in four stages. In these stages, caudal translation was performed first, followed by anterior translation, then mediolateral translation, and finally ventro-caudal translation. The procedures were performed twice a week for six weeks. The applications lasted an average of 30 minutes.
  Interventions: Other: exercises
- Control group (Experimental): A second assessment was conducted six weeks after the first assessment. No treatment w
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises — manuel therapy and exercises

SUMMARY:
This study was conducted to investigate the effect of manual therapy applications on pain, range of motion and joint position sense in individuals with rheumatoid arthritis who have temporomandibular joint dysfunction. The 57 patients included in the study were divided into 3 groups by simple randomization. Group 1 received myofascial mobilization of masticatory muscles and group 2 received temporomandibular joint mobilization twice a week for 6 weeks. The control group received no treatment. The groups were evaluated twice, before and after treatment. The control group underwent a second evaluation 6 weeks after the first evaluation. C-ROM was used to evaluate cervical range of motion and joint position sensation, millimeter ruler was used to evaluate TMJ range of motion, Algometer was used to evaluate pressure pain threshold of muscles, Headache Impact Test-HIT-6 was used for headache, Fonseca Anamnestic Index (FAI) and Jaw Function Limitation Scale-20 (JFLS-20) were used for temporomandibular dysfunction severity, Generalized Anxiety Disorder-7 was used for emotional state. In the cervical range of motion, the myofascial group showed significant normal range of motion improvements only in the flexion and lateral flexion directions, while no benefit was obtained in the extension and rotation directions. In the joint mobilization group, significant improvements were observed in all directions (flexion, extension, lateral flexion, rotation) (p<0.05). In the evaluation of cervical joint position sensation, improvements in joint position sensation were observed in all directions in the joint mobilization group. In the myofascial mobilization group, limited improvements were observed in some directions, but most of the variables decreased (p<0.05). In the measurement of pressure pain thresholds, a decrease was observed in the two treatment groups before and after treatment and compared to the control group (p<0.05), while no statistically significant difference was detected in any variable in the comparison between the treatment groups (P>0.05). Patients in the two treatment groups showed an increase in mandibular range of motion in all directions compared to both the pre- and post-treatment and control groups (p<0.05), while no statistically significant difference was detected in any variable in the comparison between the treatment groups (P>0.05). Joint mobilization and myofascial mobilization applications significantly reduced headache, anxiety severity and improved jaw function. There was a significant decrease in HIT-6, GAD-7, JFLS-20 total, JFLS-20 mastication, JFLS-20 mobility, JFLS-20 communication and Fonseca scores in both groups (p<0.05), while no statistically significant difference was found in any variable in the comparison of treatment groups (P>0.05). It was observed that myofascial mobilization and joint mobilization applications had positive effects on pain, mandibular range of motion, cervical joint range of motion and joint position sensation, jaw functions, headache and anxiety level in individuals with rheumatoid arthritis with temporomandibular joint dysfunction.

DETAILED DESCRIPTION:
This study was conducted to investigate the effect of manual therapy applications on pain, range of motion and joint position sense in individuals with rheumatoid arthritis who have temporomandibular joint dysfunction. The 57 patients included in the study were divided into 3 groups by simple randomization. Group 1 received myofascial mobilization of masticatory muscles and group 2 received temporomandibular joint mobilization twice a week for 6 weeks. The control group received no treatment. The groups were evaluated twice, before and after treatment. The control group underwent a second evaluation 6 weeks after the first evaluation. C-ROM was used to evaluate cervical range of motion and joint position sensation, millimeter ruler was used to evaluate TMJ range of motion, Algometer was used to evaluate pressure pain threshold of muscles, Headache Impact Test-HIT-6 was used for headache, Fonseca Anamnestic Index (FAI) and Jaw Function Limitation Scale-20 (JFLS-20) were used for temporomandibular dysfunction severity, Generalized Anxiety Disorder-7 was used for emotional state. In the cervical range of motion, the myofascial group showed significant normal range of motion improvements only in the flexion and lateral flexion directions, while no benefit was obtained in the extension and rotation directions. In the joint mobilization group, significant improvements were observed in all directions (flexion, extension, lateral flexion, rotation) (p<0.05). In the evaluation of cervical joint position sensation, improvements in joint position sensation were observed in all directions in the joint mobilization group. In the myofascial mobilization group, limited improvements were observed in some directions, but most of the variables decreased (p<0.05). In the measurement of pressure pain thresholds, a decrease was observed in the two treatment groups before and after treatment and compared to the control group (p<0.05), while no statistically significant difference was detected in any variable in the comparison between the treatment groups (P>0.05). Patients in the two treatment groups showed an increase in mandibular range of motion in all directions compared to both the pre- and post-treatment and control groups (p<0.05), while no statistically significant difference was detected in any variable in the comparison between the treatment groups (P>0.05). Joint mobilization and myofascial mobilization applications significantly reduced headache, anxiety severity and improved jaw function. There was a significant decrease in HIT-6, GAD-7, JFLS-20 total, JFLS-20 mastication, JFLS-20 mobility, JFLS-20 communication and Fonseca scores in both groups (p<0.05), while no statistically significant difference was found in any variable in the comparison of treatment groups (P>0.05). It was observed that myofascial mobilization and joint mobilization applications had positive effects on pain, mandibular range of motion, cervical joint range of motion and joint position sensation, jaw functions, headache and anxiety level in individuals with rheumatoid arthritis with temporomandibular joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 18 and 65
* Have been diagnosed with rheumatoid arthritis according to the ACR/EULAR 2010 criteria
* Be in the chronic phase of the disease
* Have temporomandibular joint dysfunction according to the RDC/TMD criteria
* Have intact cognitive functions
* Individuals who agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* - Maksillofasiyal travma ve cerrahi öyküsü olanlar
* Son 6 ayda ortodontik tedavi öyküsü olanlar
* Trigeminal nevralji ve/veya fasiyal sinir paralizisi öyküsü olanlar
* Romatoid Artrit dışında ek bir romatolojik hastalığı olanlar
* Ağız içi splint kullanıyor olmak
* Protez diş kullanımı ve molar dişlerde eksiklik
* Servikal bölgeye ve temporomandibular eklem disfonksiyonuna yönelik son 6 ayda Manuel - Terapi, enjeksiyon vb. benzeri tedavi görmüş olmak

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
assessing cervical joint range of motion and joint position sense | 6 weeks
  c-rom
TME Movement Clarity, | 6 weeks
  Millimetre Ruler
pressure pain threshold of muscles | 6 weeks
  Algometer
headache | 6 weeks
  Headache Impact Test- HIT-6
Severity of temporomandibular dysfunction | 6 weeks
  Fonseca Anamnestik İndeksi ve Çene Fonksiyon Kısıtlanma Skalası-20(JFLS-20),

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko Unıversıty, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No